CLINICAL TRIAL: NCT01929278
Title: A Single-Center, Evaluator-Blinded, Randomized, Placebo Controlled, Phase 1 Clinical Trial Evaluating The Phototoxic Potential Of Topically Applied Clindamycin 1.0% - Tretinoin 0.025% Gel (Ct Gel) In Healthy Volunteers
Brief Title: W0265-103: A Single-Center, Evaluator-Blinded, Randomized, Placebo Controlled, Phase 1 Clinical Trial Evaluating The Phototoxic Potential Of Topically Applied Clindamycin 1.0% - Tretinoin 0.025% Gel (Ct Gel) In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 114729
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CT Gel patch (Experimental): CT Gel is a reformulation of VELAC Gel that contains the same active ingredients (clindamycin 1% and tretinoin 0.025%) in a modified vehicle. The test article was placed on a separate occlusive patch at volumes of 200 µL per patch.
  Interventions: Drug: CT Gel (clindamycin 1% and tretinoin 0.025%)
- Vehicle gel patch (Placebo Comparator): The test article was placed on a separate occlusive patch at volumes of 200 µL per patch.
  Interventions: Other: Vehicle gel patch
- Blank patch (Experimental): Blank patches did not contain CT Gel or vehicle gel.
  Interventions: Other: Blank patch

INTERVENTIONS:
Drug: CT Gel (clindamycin 1% and tretinoin 0.025%) — Three CT Gel patches were concurrently applied to designated test sites by trained technicians and held in place with hypoallergenic tape. Patches were prepared no longer than 30 minutes prior to application to study subjects. A minimum distance of ¾ of an inch from patch pad to patch pad was maintained on a subject's back. Approximately 24 ±1 hours after patch application, test patches were removed by trained technicians. Patch sites were evaluated for signs of inflammation according to procedures.
  Arms: CT Gel patch
Other: Vehicle gel patch — Three vehicle gel patches were concurrently applied to designated test sites by trained technicians and held in place with hypoallergenic tape. Patches were prepared no longer than 30 minutes prior to application to study subjects. A minimum distance of ¾ of an inch from patch pad to patch pad was maintained on a subject's back. Approximately 24 ±1 hours after patch application, test patches were removed by trained technicians. Patch sites were evaluated for signs of inflammation according to procedures. 2. Vehicle gel contained the identical ingredients and packaging as CT Gel but without the active ingredients. All vehicle gel used during the study was from batch ZLU C.
  Arms: Vehicle gel patch
Other: Blank patch — Three blank patches were concurrently applied to designated test sites by trained technicians and held in place with hypoallergenic tape. Patches were prepared no longer than 30 minutes prior to application to study subjects. A minimum distance of ¾ of an inch from patch pad to patch pad was maintained on a subject's back. Approximately 24 ±1 hours after patch application, test patches were removed by trained technicians. Patch sites were evaluated for signs of inflammation according to procedures. 3. Occlusive patches consisted of a non-woven cotton pad (Webril [approximately 2 cm x 2 cm]) covered and secured on all sides by an occlusive hypoallergenic tape (approximately 4 cm x 4 cm).
  Arms: Blank patch

SUMMARY:
Clindamycin 1.0% - tretinoin 0.025% gel (CT Gel) is a reformulation of VELAC Gel that contains the same active ingredients (clindamycin 1.0% and tretinoin 0.025%) in a modified vehicle. This was a single-center, evaluator-blinded, randomized, placebo (vehicle)-controlled phase 1 study to evaluate the phototoxic potential of CT Gel using 24 hour single applications of 3 sets of 3 study patches. The study expected to enroll approximately 40 healthy adult volunteers. Each set of study patches consisted of a CT Gel patch, a vehicle gel patch, and a blank patch (did not contain CT Gel or vehicle gel).

After concurrent 24-hour single applications of all 9 patches, 1 set of patches (set A) was removed, and those sites were irradiated with 16 joules/cm2 of ultraviolet A light (UVA) and 0.75 minimal erythema dose (MED) with UVA/ultraviolet B light (UVB). The second set of patches (set B) was removed, and those sites were irradiated with 16 joules/cm2 of UVA, 0.75 MED with UVB/UVA, followed by 15 joules/cm2 of visible light (VIS). The third set of patches (set C) was then removed, and those sites served as a non irradiated control. Inflammatory responses and other cutaneous effects were scored 1 hour after patch removal and during follow-up visits at 24, 48, and 72 hours after patch removal.

ELIGIBILITY:
Inclusion Criteria:

1. The capability of understanding and providing signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol-specific procedures were performed.
2. Male or female subjects aged from 18 to 65 years, inclusive, at time of consent.
3. The ability to complete the study and to comply with study instructions.
4. Possessed Fitzpatrick skin type I (always burns easily; never tans), II (always burns easily; tans minimally), or III (burns moderately; tans gradually) that would not interfere with the reading of any skin responses. Determination of skin types was based on sunburn and tanning histories, as well as subjects' opinions of their responses to the first 30 to 45 minutes of sun exposure.
5. Sexually active females of childbearing potential who agreed to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential was defined as one who was biologically capable of becoming pregnant, including perimenopausal women who were less than 2 years from their last menses. Acceptable contraceptive methods included the following:

   * Hormonal contraception, including oral, injectable, or implantable methods started at least 2 months prior to screening. If hormonal contraception was started less than 2 months prior to screening, then a form of non-hormonal contraception was to have been added until the third continuous month of hormonal contraception was completed.
   * Two forms of non hormonal contraception, including intrauterine devices or properly used barrier methods (eg, male or female condoms, diaphragm, or cervical cap). Subjects with surgical sterilization, including tubal ligation or partner's vasectomy, were to have used a form of non-hormonal contraception. A barrier method or sterilization plus spermatocide were acceptable.

Women who were not currently sexually active or lactating agreed to use a medically accepted method of contraception if she became sexually active while participating in the study.

Exclusion Criteria:

1. Currently diagnosed with cancer or had a previous history of cancer, including skin cancer, or severe photodamaged skin. Severe photodamaged skin was characterized by yellow-gray color, wrinkles with no visible normal skin, and prior skin malignancies.
2. Female subjects who were pregnant, attempting to become pregnant, or breast feeding.
3. Received any investigational drug within 4 weeks of study day 1 or who were scheduled to receive an investigational drug other than the study product during the study.
4. Used contraindicated prescription drugs within 4 weeks or 5 half-lives, whichever was longer, of first dose of study product, unless agreed as not clinically relevant by the principal investigator and the project physician.
5. Participated in a previous study of the same study product.
6. Current use of any medication which, in the opinion of the investigator, may have affected the evaluation of the study product or placed the subject at undue risk.
7. Suffered from any disease or condition which, in the opinion of the investigator, may have affected the evaluation of the study product or placed the subject at undue risk.
8. Any major illness within 30 days before the screening examination.
9. Considered immunocompromised or using immunosuppressant drugs.
10. Clinically relevant history of or current evidence of abuse of alcohol or other drugs.
11. History of known or suspected intolerance to any of the ingredients of the study products (ie, test and comparator products), to the hypoallergenic tape, or to the cotton patches.
12. Clinically relevant history or presence of respiratory (including chronic asthma requiring repetitive drug interventions), gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, or connective tissue diseases or disorders.
13. Considered unable or unlikely to attend the necessary visits.
14. History of severe reactions from exposure to sunlight, including previous experience with photoallergy, solar urticaria, polymorphous light eruptions, or other photo exacerbated systemic diseases.
15. Current use or expected use of photosensitizing medications (over-the-counter and prescription), herbal supplements, or any use of a known photosensitizing material.
16. Clinically significant skin diseases contraindicating participation or interfering with test site evaluations, including psoriasis, eczema, atopic dermatitis, acne, dysplastic nevi, or other skin pathologies.
17. Investigator inability to evaluate the skin in and around the potential test sites due to sunburns, unevenness in skin tones, tattoos, scars, excessive hair, freckles, birthmarks, moles, or other skin abnormalities.
18. Used topical medications (eg, corticosteroids or immunosuppressives) on potential test sites within the last 7 days prior to screening visit 1.
19. Currently receiving allergy injections, or due to receive an injection, within 7 days prior to screening visit 1, or expected to begin injections during study participation.
20. Used antihistamines or prescription anti inflammatory drugs within 72 hours of the day 1 visit. Permitted exceptions were acetaminophen at recommended doses and aspirin at doses of ≤81 mg/day.
21. Participated in any patch test study for irritation or sensitization or any test involving ultraviolet exposures within the last 4 weeks.
22. Employees of Hill Top Research or Stiefel Laboratories involved in the study, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee involved in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-12-08 (Actual); Primary Completion 2008-12-19 (Actual); Study Completion 2008-12-19 (Actual)

PRIMARY OUTCOMES:
Inflammatory responses (erythema and local skin reactions) or superficial effects (if observed) will be scored according to the erythema, local skin reaction, and superficial effects grading scales. | 6 - 11 days
  In cases where the patch area is larger than the irradiated area, only the irradiated areas will be scored unless reactions outside the irradiated area exhibit unusual responses. Scores represent the presence of clinically significant effects on at least 25% of the test site. Questionable, barely perceptible, or minimal reactions involving less than 25% of the test site will not be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: Results for study 114729 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114729?search=study&search_terms=114729#rs